CLINICAL TRIAL: NCT03935113
Title: Effects of Kinesio Taping for Upper Limb Function of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N201811021
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2019-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KT group (Experimental): The paretic upper limb is a common consequence of stroke that increases activity limitation.
  Interventions: Other: Kinesio taping

INTERVENTIONS:
Other: Kinesio taping — In KT group, KT was applied using the insertion-origin muscle and space-correction technique of affected upper limb with stroke patients.

SUMMARY:
Patients with stroke in the brain, due to central nervous system damage, lack of correct action patterns, limited joint movement of upper limbs, affecting the patient's performance. The Kinesio taping effect is to facilitate the muscle activity of upper limb. This program is intended to provide a treatment for patients with chronic stroke, and to observe their upper limb movements before and after using the Kinesio taping.

DETAILED DESCRIPTION:
Motor impairment is the main cause of disability after stroke, leading to major health problems. Research has shown that the most common consequence of stroke is the paresis of limbs.The ability to live independently after a stroke depends on the recovery of motor functions,particularly those of the upper limb.The core concept of the Kinesio taping is to influence the brain through the sensory input, stimulate the nervous system, and improve the motor performance of the stroke patient.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke hemiplegia, at least 6 months since onset
* Ability to communicate and understand instructions.

Exclusion Criteria:

* Skin problems, wounds, or infection on the affected upper limb.
* The experience of using the Kinesio taping.
* A history of allergy tothe Kinesio taping.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) from pre to post-intervention. | up to 30 minutes.
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
Change in Action Research Arm Test (ARAT) from pre to post-intervention. | up to 30 minutes.
  The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among post-stroke hemiplegia.
Change in Box and Block Test (BBT) from pre to post-intervention. | up to 30 minutes.
  The Box and Block Test (BBT) measures unilateral gross manual dexterity for stroke patients.

SECONDARY OUTCOMES:
Change in Motor Activity Log (MAL) from pre to post-intervention. | up to 20 minutes.
  The Motor Activity Log (MAL) is a semi-structured interview to assess arm function.

CONTACTS AND LOCATIONS:
Locations (1):
- Wang Fang hospital, Taipei, Taipei City, Taiwan